CLINICAL TRIAL: NCT06809465
Title: Effect of Supplementation of Probiotic Bifidobacterium Bifidum PRL2010) in Pregnancy for the Prevention of Atopic Dermatitis in Children: A Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Probiotic Bifidobacterium Bifidum PRL 2010 in the Prevention of Atopic Dermatitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ref. 6205/Sapienza University
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Bifidobacterium bifidum PRL2010 (Bactopral®) (Experimental): Participants in this arm will receive probiotic Bifidobacterium bifidum PRL2010 (Bactopral®) supplement. Each Bactopral®s sachet contains 1 billion CFU/sachet of the Bifidobacterium bifidum PRL2010. Mothers will take one sachet daily starting at the 36th week of pregnancy and continuing until delivery. During the first two months postpartum, mothers will continue daily doses. Infants will then receive the same probiotic from the 3rd to 6th month of life. Probiotic powder will be mixed with breast milk and administered via teaspoon or syringe.
  Interventions: Dietary Supplement: Bactopral®
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo identical in appearance, smell, and taste to the probiotic. The placebo contains bacteria-free maltodextrins. Administration will follow the same schedule as the probiotic arm.
  Interventions: Other: Plcebo

INTERVENTIONS:
Dietary Supplement: Bactopral® — Oral Probiotic Bifidobacterium bifidum PRL2010 supplement
  Arms: Probiotic Bifidobacterium bifidum PRL2010 (Bactopral®)
Other: Plcebo — Oral placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of supplementation with Bifidobacterium bifidum PRL2010 during pregnancy in preventing atopic dermatitis in children. Pregnant women with a history of atopy or family history of allergies will be randomized to receive either the probiotic or a placebo. Outcomes include the incidence and severity of atopic dermatitis in infants up to 12 months of age.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a growing public health concern due to its increasing prevalence and significant impact on quality of life. This randomized, double-blind, placebo-controlled pilot study investigates the efficacy of Bifidobacterium bifidum PRL2010 in preventing AD when administered during pregnancy. Women aged 18-45 with a history of atopy or family history of allergies will be recruited and randomized into two groups: one receiving the probiotic and the other receiving a placebo. The intervention will begin at the 36th week of pregnancy and continue postpartum during breastfeeding for two months. Infants will subsequently receive the same treatment from the 3rd to 6th month of life. Outcomes include the presence and severity of AD assessed using the SCORAD index and additional allergy tests at 3, 6, and 12 months of age. This pilot aims to assess feasibility, safety, and initial efficacy data for future larger-scale studies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-45 years.
* Presence of allergic manifestations or a positive family history of allergies.
* Normal pregnancy without complications (e.g., no risk of eclampsia or gestational diabetes).
* Residing in Rome.
* Non-smoker and non-smoking partner.
* Absence of pets.
* Planning natural childbirth.
* Intention to breastfeed for at least 3 months.

Exclusion Criteria:

* Complications during pregnancy (e.g., preterm birth before 36 weeks).
* Infants with necrotizing enterocolitis or congenital, chronic, or metabolic diseases.
* Immunodeficiencies in mother or child.
* Failure to meet any inclusion criteria during the study period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is limited to pregnant women as it investigates the effect of Bifidobacterium bifidum PRL2010 supplementation during pregnancy on the prevention of atopic dermatitis in their infants.
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Atopic Dermatitis in Infants | 12 months from birth
  The presence of atopic dermatitis in infants will be evaluated using the SCORAD index at 3, 6, and 12 months of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Department of Maternal Infantile and Urological Sciences, Division of Pediatric Allergology and Immunology, Roma, Italy

IPD SHARING:
Plan to Share IPD: No